CLINICAL TRIAL: NCT00287573
Title: A Prospective, Randomized Trial Evaluating Slow-Release Formulation TAXUS Paclitaxel-Eluting Coronary Stent in the Treatment of In-Stent Restenosis
Brief Title: Randomized Trial Evaluating Slow-Release Formulation TAXUS Paclitaxel-Eluting Coronary Stent in the Treatment of In-Stent Restenosis
Acronym: TAXUS V ISR
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Marcie Clarkin, Boston Scientific
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: S5442; TAXUS V ISR
Record Dates: First submitted 2006-02-03; First posted 2006-02-07 (Estimated); Last update posted 2010-08-06 (Estimated); Status verified 2010-08

CONDITIONS: Coronary Restenosis
MeSH Terms: conditions — Coronary Restenosis | interventions — Brachytherapy

ARMS (2):
- Arm 1 (Experimental)
  Interventions: Device: TAXUS Express2
- Arm 2 (Active Comparator)
  Interventions: Procedure: Brachytherapy (beta source)

INTERVENTIONS:
Device: TAXUS Express2 — Paclitaxel-Eluting Coronary Stent System
  Arms: Arm 1
Procedure: Brachytherapy (beta source) — Brachytherapy (beta source)
  Arms: Arm 2

SUMMARY:
The objective of this study is to evaluate the safety and effectiveness of the TAXUS Express2 Paclitaxel-Eluting Coronary Stent System as compared to brachytherapy in patients experiencing in-stent restenosis.

DETAILED DESCRIPTION:
Percutaneous approaches to in-stent restenosis (ISR) have included balloon angioplasty alone, rotational atherectomy, cutting balloon angioplasty, directional coronary atherectomy, excimer laser angioplasty, placement of a second stent or any combination thereof, and intra-coronary brachytherapy. Of these, only brachytherapy has been shown to reduce recurrent restenosis after PCI for ISR, - and is now considered the standard of care. Logistical considerations in establishing and maintaining a radiation program have limited the widespread availability of this modality. These considerations include the need for involvement of radiation oncologists, physicists, and safety officers; nuclear licensing requirements; need for increased shielding and safety training; equipment and procedural complexities; as well as increased procedural time and costs. Furthermore, recurrent ISR after brachytherapy may still occur. Stent based drug delivery for the treatment of ISR holds promise as a much simpler, safer and potentially more effective alternative to brachytherapy.

This is a prospective, randomized (1:1), open-label, multicenter, safety and efficacy trial for the treatment of in-stent restenosis. The primary objective is to demonstrate a superior or non-inferior 9-month target vessel revascularization (TVR) rate for TAXUS-SR stent compared to intra-coronary brachytherapy (beta source).

ELIGIBILITY:
Inclusion Criteria:

* Cumulative target lesion length is </= 46 mm (visual estimate).
* Reference vessel diameter (RVD) is >/= 2.5 and </= 3.75 mm (visual estimate)
* Left ventricular ejection fraction (LVEF) is >/= 25%

Exclusion Criteria:

* Any previous or planned treatment with a non-study anti-restenotic drug-coated or drug-eluting coronary stent in the target vessel. (Note:previous or planned treatment with heparin or phosphorylcholine coated stents is acceptable, as long as, the procedure with the non-study stent meets the protocol defined criteria for non-target lesion interventions.)
* Previous or planned treatment with intra-coronary brachytherapy (gamma or beta source) in the target vessel
* Previous external radiotherapy to the heart or target vessel area
* Known genetic radiation sensitivity disorders (i.e. ataxia-telangiectasia, etc.)
* Side branch of the target lesion includes ostial narrowing >/= 50% diameter stenosis (DS) and is >/= 2.0 mm diameter
* Target lesion has been previously treated for ISR with the placement of a second stent(s), which covers >/= 50% of the original stent length (a true "stent sandwich")
* Target vessel is pre-treated with an unapproved device, directional or rotational coronary atherectomy, laser, or transluminal extraction catheter immediately prior to delivery of randomized treatment (stent placement or intra-coronary brachytherapy)
* Recent myocardial infarction (MI) (symptom onset </= 72 hours prior to randomization)
* CK-MB >2x the local laboratory's upper limit of normal (ULN) (refers to a measured value on the day of the index procedure as drawn per protocol)
* Anticipated treatment with warfarin during any period in the 6 months post index procedure
* Anticipated treatment with paclitaxel, oral rapamycin or colchicine during any period in the 9 months post index procedure
* Planned use of both the study stent and a non-study stent (i.e., commercial stent) in the treatment of the target lesion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 488 (Actual)
Dates: Start 2003-06; Primary Completion 2004-12 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
Rate of Target Vessel Revascularization | 9 Months

SECONDARY OUTCOMES:
Incidence of composite major adverse cardiac events (MACE) and the individual components of MACE | assessed at discharge, 1, 4 and 9 months post index procedure and annually for 5 years
Stent thrombosis rate | 5 Years
Target Vessel Failure (TVF, defined as any ischemia-driven revascularization of the target vessel, MI related to the target vessel, or death related to the target vessel). | 5 Years
Clinical procedural success and technical success | 5 Years
Binary restenosis rate | 5 years
Evaluate outcomes and treatment of recurrent restenosis in the TAXUS stent arm | 5 Years
Absolute lesion length | 9 Months
Reference Vessel Diameter (RVD) | 9 Months
Minimum Lumen Diameter (MLD) | 9 Months
Percent diameter stenosis (% DS) | 9 Months
Acute gain | 9 Months
Late loss | 9 Months
Loss index | 9 Months
Patterns of recurrent restenosis, including edge effect | 9 Months
Coronary aneurysm | 9 Months
Identification of potential safety issues. | 9 Months
Change in neointimal volume from post procedure to follow-up | 9 Months
Change in MLD within the stent or area of brachytherapy | 9 Months
Minimum lumen area (MLA) within the stent or area of brachytherapy | 9 Months
Lumen, plaque and vessel measurements at the treatment edges (outside of the stent or area of brachytherapy) | 9 Months

CONTACTS AND LOCATIONS:
Overall Officials: Gregg W. Stone, MD, Principal Investigator — Columbia University; Stephen G. Ellis, MD, Principal Investigator — The Cleveland Clinic
Locations (42):
- United States (40):
  - Baptist Medical Center Princeton, Birmingham, Alabama
  - Scripps Green Hospital, La Jolla, California
  - Mercy General Hospital, Sacramento, California
  - Stanford Medical Center, Stanford, California
  - Aurora Denver Cardiology, Aurora, Colorado
  - Washington Hospital Center, Washington D.C., District of Columbia
  - Florida Hospital, Orlando, Florida
  - Piedmont Hospital, Atlanta, Georgia
  - Ochsner Clinic Foundation, New Orleans, Louisiana
  - Maine Medical Center, Portland, Maine
  - Washington Adventist Hospital, Takoma Park, Maryland
  - Tufts Medical Center, Boston, Massachusetts
  - Lahey Clinic Hospital, Burlington, Massachusetts
  - University of Massachusetts Memorial Medical Center, Worcester, Massachusetts
  - Spectrum Health Hospitals, Grand Rapids, Michigan
  - Cardiac & Vascular Research Center of Northern Michigan, Petoskey, Michigan
  - Abbott Northwestern Hospital, Minneapolis, Minnesota
  - Saint Luke's Hospital, Kansas City, Missouri
  - Barnes Jewish Hospital, St Louis, Missouri
  - Nebraska Heart Institute, Lincoln, Nebraska
  - Albany Medical Center/Capital Cardiovascular Associates, Albany, New York
  - Buffalo General Hospital, Buffalo, New York
  - Columbia University Medical Center, New York, New York
  - Lenox Hill Hospital, New York, New York
  - Mid-Carolina Cardiology Research Division/Presbyterian Hospital, Charlotte, North Carolina
  - LeBauer Cardiovascular Research Foundation, Greensboro, North Carolina
  - Forsyth Medical Center, Winston-Salem, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - The Lindner Clinical Trial Center, Cincinnati, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - North Ohio Research, Ltd, Elyria, Ohio
  - Oklahoma Cardiovascular Research Group, Oklahoma City, Oklahoma
  - St. Mary's Medical Center, Langhorne, Pennsylvania
  - The Miriam Hospital, Providence, Rhode Island
  - South Carolina Heart Center, Columbia, South Carolina
  - St. Thomas Hospital, Nashville, Tennessee
  - South Austin Hospital/Capital Cardiovascular Specialists, Austin, Texas
  - The Methodist Hospital Research Institute in Cardiovascular Interventions, Houston, Texas
  - University of Virginia, Charlottesville, Virginia
  - Swedish Medical Center, Seattle, Washington
- Canada (2):
  - Sunnybrook & Women's College Health Sciences Centre, Toronto, Ontario
  - Toronto General Hospital, Toronto, Ontario

REFERENCES:
- [Result] Stone GW, Ellis SG, O'Shaughnessy CD, Martin SL, Satler L, McGarry T, Turco MA, Kereiakes DJ, Kelley L, Popma JJ, Russell ME; TAXUS V ISR Investigators. Paclitaxel-eluting stents vs vascular brachytherapy for in-stent restenosis within bare-metal stents: the TAXUS V ISR randomized trial. JAMA. 2006 Mar 15;295(11):1253-63. doi: 10.1001/jama.295.11.1253. Epub 2006 Mar 12. PMID 16531618